CLINICAL TRIAL: NCT00598780
Title: Long-term Evaluation of Safety and Treatment Satisfaction With Levocetirizine in Routine Clinical Practice in the Czech and Slovak Republics - Non-interventional Study
Brief Title: Evaluation of Safety of Levocetirizine in Routine Clinical Practice-non- Interventional Study
Status: Completed | Type: Observational
Sponsor: UCB Pharma (Industry)
Responsible Party: Sponsor
Other Study IDs: A00421
Record Dates: First submitted 2008-01-11; First posted 2008-01-23 (Estimated); Last update posted 2012-05-28 (Estimated); Status verified 2008-10

CONDITIONS: Rhinitis Allergic, Persistent
Keywords: Levocetirizine; Xyzal; Rhinitis allergic persistent; Rhinitis nonseasonal
MeSH Terms: conditions — Rhinitis, Allergic, Perennial

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: Patients with newly diagnosed persistent allergic rhinitis, within the approved age limits.

SUMMARY:
To evaluate over a period of 6 months the safety and the treatment satisfaction of newly prescribed levocetirizine in patients of age ≥ 2 years with persistent allergic rhinitis.

DETAILED DESCRIPTION:
This is a non-interventional, prospective, post-authorization, multi-centre cohort study in patients treated with levocetirizine.

The baseline data will be collected at the visit to the physician when levocetirizine is prescribed for the first time for the patient for Persistent Allergic Rhinitis. The data will then be collected during 2 visits occurring within the first 6 months of treatment, as usually scheduled in normal clinical practice in the Czech and Slovak Republics. This is after approximately 4 weeks and 6 months of treatment or earlier, if the treatment is stopped

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of persistent allergic rhinitis
* first prescription of levocetirizine for this diagnosis for this patient
* age ≥ 2 years

Exclusion Criteria:

* indications other than those defined in inclusion criteria
* history of allergic or anaphylactic reactions to levocetirizine or other derivatives and excipients included

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with newly diagnosed persistent allergic rhinitis, within the approved age limits.
  Age ≥ 2 years
Sampling Method: Probability Sample
Enrollment: 7870 (Actual)
Dates: Start 2007-09; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
Number of patients with adverse events Number and type of serious adverse events Number of patients withdrawing levocetirizine treatment due to adverse events | Six Months

SECONDARY OUTCOMES:
To evaluate the global clinical improvement on levocetirizine compared to baseline at each follow up visit. | Six months
To evaluate the treating physician's perception of patient satisfaction of levocetirizine tolerability at each follow up visit | six months
To evaluate symptoms (nasal pruritus, rhinorrhea, nasal congestion, sneezing, ocular pruritus) at each follow up visit | six months
To evaluate the impact of co-morbidities (asthma, urticaria and inflammation of upper airways) at each follow up visit | six months
To evaluate the treating physician's perception of patient satisfaction of treatment regimen effectiveness at each follow up visit | six months
To evaluate the treating physician's prescription practice in the treatment of Persistent Allergic Rhinitis | six months
To evaluate concomitant medications prescribed with levocetirizine at each follow up visit | six months
The evaluate reason for discontinuation at last follow up visit | six months
To evaluate the overall physician´s treatment satisfaction in comparison with previously used antihistamines in patient population previously treated by antihistamines at last follow up visit | six months
To evaluate the dose prescribed by the treating physician at each follow up visit | six months

CONTACTS AND LOCATIONS:
Overall Officials: UCB Clinical Trial Call Center, Study Director — +1 877 822 9493 (UCB)
Locations (1):
- UCB Pharma, Smyrna, Georgia, United States